CLINICAL TRIAL: NCT05679414
Title: Prevalence of Thrombophilic Gene Polymorphism (MTHFR C677T) in Egyptian Patients With COVID-19
Brief Title: Prevalence of Thrombophilic Gene Polymorphism (MTHFR C677T) in COVID-19patients
Acronym: (MTHFR)C677T
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Eman Badawy AbdelFattah, Associate professor of Pulmonary Medicine, Ain Shams University
Other Study IDs: FMASU R 130/2022
Record Dates: First submitted 2023-01-09; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: COVID 19 Associated Coagulopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Covid 19 patients in which MTHFR C677T genotypes was determined by RT- PCR of 2 ml EDTA blood sample.Follow up patient for 28 days as regard development of vascular thrombotic manifestation
  Interventions: Diagnostic Test: RT- PCR of 2 ml EDTA blood sample to determine MTHFR C677T genotypes
- Control group: Healthy subjects in which MTHFR C677T genotypes was determined by RT- PCR of 2 ml EDTA blood sample.
  Interventions: Diagnostic Test: RT- PCR of 2 ml EDTA blood sample to determine MTHFR C677T genotypes

INTERVENTIONS:
Diagnostic Test: RT- PCR of 2 ml EDTA blood sample to determine MTHFR C677T genotypes — Venous blood sample

SUMMARY:
Aim of the study is to find the prevalence of thrombophilic gene methylene tetrahydrofolate reductase (MTHFR) gene polymorphism in a sample of COVID-19 patients, aiming at early detection of MTHFR mutant patients and guiding preventive therapy.

DETAILED DESCRIPTION:
The inflammatory component of severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) creates a prothrombotic state that necessitates a thrombophylactic strategy for hospitalized patients. Such strategies are difficult to be standardized because certain individuals can have prothrombotic conditions, such as inherited thrombophilia, which predispose them to an additional coagulative risk. Whether outside the hospital or when admitted, patients with inherited thrombophilia need special anticoagulant attention. Identifying such patients, especially in susceptible populations like the Egyptian people, will aid primary providers in risk stratification for choosing the optimal anticoagulation plan. Case-control study which will be conducted on 33 patients who had been diagnosed as COVID-19 at Ain-Shams University isolation Hospitals and 13 healthy controls. Patients will be subjected to: Thorough history taking, Thorough clinical assessment,COVID-19 PCR+/- radiological data collection, Assessment of MTHFR C677T genotypes were determined by RT- PCR of 2 ml EDTA blood sample, Follow up patient for 28 days as regard development of vascular thrombotic manifestation (D. dimer, LL duplex, or CT chest with Pulmonary angiography if needed).

ELIGIBILITY:
Inclusion Criteria:

* All adult patients diagnosed as COVID -19 by RT-PCR will be included

Exclusion Criteria:

* Patients younger than 18 years old Patients on Antithrombotic treatment before COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed as COVID -19 by RT-PCR
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
development of vascular thrombotic manifestation | 4 weeks
  Level of D. dimer, Lower Limb duplex, or CT chest with Puplomary Angiography if needed.

CONTACTS AND LOCATIONS:
Overall Officials: Eman B AbdelFattah, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication maybe shared
Supporting Information: Study Protocol, SAP
Time Frame: 3 months after publication
Access Criteria: Through the primary investigator e-mail to other interested researchers